CLINICAL TRIAL: NCT01823614
Title: Epidemiological Study of the Co-receptor Tropism of HIV-1 Subtype A Spread in the Russian Federation Among naïve and ART-experienced Patients Using V3-based Genotyping Tools
Brief Title: Co-receptor Tropism Determination of HIV-1 Subtype A Spread in the Russian Federation Using V3-based Genotyping Tools
Acronym: CoTrAST
Status: Completed | Type: Observational
Sponsor: Dmitry Kireev (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Dmitry Kireev, scientific researcher, Central Institute of Epidemiology, Moscow, Russia
Organization: Central Institute of Epidemiology, Moscow, Russia (Other)
Other Study IDs: WS2041679
Record Dates: First submitted 2013-03-30; First posted 2013-04-04 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infection
Keywords: HIV infection; tropism determination; genotypic methodic; R5-tropic variant; X4-tropic variant
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Naïve patients, >500: The group contains patients who have not any ARV therapy experience and the level of CD4 count is more than 500 cells per mm3
- Naïve patients, 350-500: The group contains patients who have not any ARV therapy experience and the level of CD4 count is between 350 and 500 cells per mm3
- Naïve patients, <350: The group contains patients who have not any ARV therapy experience and the level of CD4 count is less than 350 cells per mm3
- ARVT <6 months: The group contains patients who have ARVT experience and obtain ART treatment less than 6 months
- ARVT from 6 months to 3 years: The group contains patients who have ARVT experience and obtain ART treatment from 6 months to 3 years
- ARVT >3 years: The group contains patients who have ARVT experience and obtain ART treatment more than 3 years

SUMMARY:
To date, all work related to the study of HIV tropism, was performed on HIV B and C subtypes. In the studied samples, HIV variants of subtype A were virtually absent. However, the existence has been shown previously of some differences in the nucleotide sequences in the V3 loop of env region of subtype A from other subtypes of virus. In the Russian Federation the subtype A of HIV-1 is predominant, and, according to some estimates, accounts for about 89% of all newly diagnosed cases of HIV infection. Thus, it seems interesting and effective to study the characteristics of HIV-1 subtype A, associated with the tropism, in the Russian Federation.

The primary objective is determination of the prevalence of R5 (chemokine receptor 5), X4 (chemokine receptor 4), and R5X4-tropic variants of HIV in HIV-infected population in Russia, and analysis of the possible features of tropism of viruses belonging to subtype A.

DETAILED DESCRIPTION:
This study is a multicenter, single-step; with estimation of the prevalence of R5, X4, and R5X4-tropic HIV variants in a population of HIV-infected Russians naïve to CCR5-antagonists antiretroviral (ARV) therapy. Additional study objectives are to identify dependence of R5- and X4-tropic HIV variants relations from the duration of infection, stage of HIV infection, the values of CD4-lymphocytes; and to compare the prevalence of R5- and X4-tropic HIV variants in cohorts of naïve and ARVT experienced patients. The study consists of single visit of all patients, during which the following procedures will be performed: obtaining of informed consent, initial evaluation of the possibility of including of the patients in the study, stratification of the patient, and if the quota for this cohort has not yet been reached, inclusion of the patient in the study. Also the detailed information will be collected on the date of birth, place of residence (region, city), date of the 1st HIV+ immune blot test, route of infection, estimation year (month) of infection, stage of HIV infection, all the known results of CD4 cell count and viral load measurements, as well as all the known schemes of ARV therapy. Additionally, the study provides a single blood sampling (of 6.4 mL volume) into a test tube in order to study the HIV tropism by sequencing. It is expected that the inclusion in the study will be completed within approximately 3 months, but this period may be extended depending on the actual inclusion of patients in each of the study centers. The Coordination Center of the study is the Central Research Institute for Epidemiology (hereinafter - the Coordination Center). Patient selection will be performed in 13 participating centers:

* The Federal Research and Methodological Center for AIDS, Moscow
* The North-West District AIDS Center, St. Petersburg
* The St. Petersburg City AIDS Center, St. Petersburg
* The Republican Clinical Hospital of Infectious Diseases, St. Petersburg
* The Volga District AIDS Center, Nizhny Novgorod
* The Republic AIDS Center of the Republic of Tatarstan, Kazan
* The Southern District AIDS Center, Rostov-on-Don
* The Ural District AIDS Center, Ekaterinburg
* The Sverdlovsk Oblast AIDS Center, Ekaterinburg
* The Yamalo-Nenets Autonomous District AIDS Center, Noyabrsk
* The Siberian Federal District AIDS Center, Omsk
* The Krasnoyarsk Regional AIDS Center, Krasnoyarsk

The study will include approximately 900 HIV-infected patients of both sexes aged 18 years or older, citizens of Russia. Patient will be selected from the AIDS centers and the Republican Clinical Hospital for Infectious Diseases, which are participants of the study. List of the study participants includes 12 AIDS centers and one Republican Clinical Infectious Diseases Hospital, so the expected number of patients will be 70 people per participant. The minimum number of patients included in the study must be at least 40 people for each participant, but the actual amount will depend on the success of patient recruitment in each of the study centers. Starting from the 4th month of study, a competitive selection of patients will be allowed, which will end as soon as the total number of enrolled patients will reach 900 people. According to the objectives of the study, HIV tropism in patients not received ART with different immune status, and experienced in ART will be analyzed, so the inclusion of patients in the study should take place according to the following quotas:

1. Naïve patients

   1. The level of CD4-lymphocytes >500 (optimum is 16 (12-18 patients))
   2. The level of CD4-lymphocytes is 350-500 (optimum is 16 (12-18 patients))
   3. The level of CD4-lymphocytes <350 (optimum is 16 (12-18 patients))
2. Patients experienced in ARV

   1. Obtains ART treatment for <6 months (optimum is 8 (4-12 patients))
   2. Obtains ARV therapy from 6 months to 3 years (optimum is 8 (4-12 patients))
   3. Obtains ART treatment for >3 years (optimum is 8 (4-12 patients)) If within 3 months after the start of the patient selection in the study it will be impossible to complete a cohort, quotas may be revised.

Scheme of the study procedures. The study procedures

* Obtaining of the informed consent
* In/exclusion criteria evaluation
* Check that the patient belongs to the cohort for which the quota is not reached
* Filling the Case Report Form for the study participant
* Blood sampling Laboratory procedures
* Determination of HIV tropism by sequencing
* Determination of HIV viral load†
* Determination of the quantity of CD4-lymphocytes† † Carried out only when the routine analysis is necessary List of estimated parameters. To study of HIV tropism by sequencing, to perform standard laboratory tests, and to determine the subtype of HIV (that is conducted by the Coordination Center selectively in 10% of the patients) blood sampling will be carried out in all patients.

Determination of HIV tropism by sequencing.

Procedure of HIV tropism determination in a sample involves the consistent implementation of the following stages: extraction of nucleic acids from the blood sample, amplification of the env gene of HIV genome, determining the nucleotide sequence of the resulting specific DNA product and its analysis by means of the Internet resource geno2pheno, located at http://coreceptor.bioinf.mpi-inf.mpg.de/index.php. According to the instructions to a set of reagents for tropism study, there are two possible results:

1. a clinical sample contains a R5-tropic virus,
2. a clinical sample contains a non-R5-tropic virus. An important additional result is the value of FPR (false positive rate), which reflects a degree of reliability of HIV tropism in a sample. Therefore, the FPR value is also presented in report containing the results of the analysis.

Standard laboratory tests. The standard laboratory tests mean measuring of viral load in a plasma sample, as well as CD4 cell count. These studies are carried out only in case when they are routinely needed. When they are performed, the results are provided in the Case Report Form of the study participant.

Determination of HIV subtype. Determination of HIV subtype is carried out by Coordination Center selectively in 10% of patients after receipt by the Coordination Center of clinical samples from all study participants (study centers). Determination of subtype includes the following stages: extraction of nucleic acids from a plasma sample, amplification of fragment of pol region of the HIV genome, determining the nucleotide sequence of obtained specific DNA products, and their bioinformatics analysis by means of Internet applications REGA Subtyping tool and Comet.

General information about the methods of statistical analysis. Parameters of descriptive statistics will be calculated for the indices for the patients and human immunodeficiency virus by calculating the proportion of patients showing some signs of corresponding categorical variables and by calculating the mean values, standard deviations, medians, 25 and 75 percentiles, minimum and maximum values of the distribution of all continuous variables from all patients with the results of their evaluation.

Also proportions of patients from different regions at different stages of the disease, and infected with HIV variants with different tropism will be calculated. Evaluation of reliability of differences of categorical variables (for example, when differences in the distribution of HIV variants with different tropism in different regions) will be performed using the chi-square test. Estimation of reliability of differences of continuous variables (eg, the level of HIV viral load) will be performed using parametric (eg, t test, ANOVA) or nonparametric (eg, Wilcoxon rank-sum test) methods.

Univariate and multivariate logistic (when the dependent variable is binary) and linear regression (when the dependent variable is continuous) analyses will be used to assess associations between exploratory (eg, CXCR4-tropic variants) and dependent (eg, the level of HIV viral load) variables.

All statistical tests will be two-sided, with 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed HIV infection
* Confirmation of informed consent provided in writing
* Russian Federation citizenship
* Age 18 years and older
* Absence of pregnancy at the time of obtaining of biological material
* Availability of data about the date of 1st positive immune blot test, date of diagnosis and formulation of the clinical diagnosis, the result of viral load analysis performed in the previous 3 months, measuring of CD4 cell count performed in the previous 3 months, information about the ongoing ARV therapy for patients receiving antiretroviral therapy

Exclusion Criteria:

* Pregnancy at the time of obtaining of biological material
* Patients receiving cytotoxic agents due to chemotherapy of cancer
* Patients receiving immunomodulatory drugs
* Participation in clinical trials with experimental drugs
* Experience of using of CCR5-antagonists
* Any condition which in the opinion of the investigator may affect the evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 943 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Kireev, PhD, Principal Investigator — Central Research Institute for Epidemiology
Locations (1):
- Central Research Institute for Epidemiology, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of patients will be conducted during 4 months of study. Patients will be selected from the AIDS centers and the Republican Clinical Hospital for Infectious Diseases, which are participants of the study. Totally there will be 12 AIDS centers. Expected number of patients will be 70 people per participant.
Pre-assignment Details: Patient exclusion criteria: Pregnancy at the time of obtaining of biological material for women, patients receiving cytotoxic agents, patients receiving immunomodulatory drugs, pParticipation in clinical trials with experimental drugs, experience of using of CCR5-antagonists.
Period: Overall Study
Arm/Group | Naïve Patients, >500 | Naïve Patients, 350-500 | Naïve Patients, <350 | ARVT <6 Months | ARVT From 6 Months to 3 Years | ARVT >3 Years
Started | 179 | 140 | 176 | 122 | 172 | 154
Completed | 179 | 140 | 176 | 122 | 172 | 154
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of naive patients should be more than number of treatment-experienced patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Naïve Patients, >500 | Naïve Patients, 350-500 | Naïve Patients, <350 | ARVT <6 Months | ARVT From 6 Months to 3 Years | ARVT >3 Years | Total
Number analyzed (Participants) | 179 | 140 | 176 | 122 | 172 | 154 | 943
Age, Continuous [Mean (Full Range); unit: years] | 32 [18 to 60] | 33 [18 to 63] | 35 [22 to 64] | 35 [18 to 65] | 36 [21 to 68] | 37 [24 to 73] | 35 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 79 | 96 | 61 | 95 | 73 | 509
  Male | 74 | 61 | 80 | 61 | 77 | 81 | 434
Nadir CD4 cell count [Median (Full Range); unit: cells/µl] | 664 (50) [501 to 1716] | 413 (50) [351 to 499] | 33 (50) [15 to 349] | 288 (50) [5 to 1276] | 350 (50) [23 to 2112] | 394 (50) [10 to 1201] | 380 (50) [5 to 2112]

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Prevalence of R5 and X4-tropic Variants of HIV in HIV-infected Population in Russia
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Naïve Patients, >500 | Naïve Patients, 350-500 | Naïve Patients, <350 | ARVT <6 Months | ARVT From 6 Months to 3 Years | ARVT >3 Years
Number analyzed (Participants) | 161 | 116 | 159 | 110 | 141 | 126
participants
  R5-tropic | 123 | 85 | 114 | 78 | 86 | 82
  X4-tropic | 38 | 31 | 45 | 32 | 55 | 44

2. Secondary Outcome: Estimation of the R5- and X4-tropic HIV Variants Ratio Stratified by CD4 Cell Count
Time Frame: 24 weeks
Measure: Number; unit: participants
Groups:
- CD4 Cell Count > 500: Group which contains patients with CD4 nadir more than 500 cell/mkl at the moment of enrollment
- CD4 Cell Count 350-500: Group which contains patients with CD4 nadir between 350 and 500 cell/mkl at the moment of enrollment
- CD4 Cell Count < 350: Group which contains patients with CD4 nadir less than 350 cell/mkl at the moment of enrollment
Arm/Group | CD4 Cell Count > 500 | CD4 Cell Count 350-500 | CD4 Cell Count < 350
Number analyzed (Participants) | 243 | 216 | 364
participants
  R5-tropic | 179 | 160 | 239
  X4-tropic | 64 | 56 | 125

3. Other Pre Specified Outcome: Estimation of the R5- and X4-tropic HIV Variants Ratio Stratified by CD4 Cell Count Among Naive Patients
Time Frame: 24 weeks
Measure: Number; unit: participants
Groups:
- CD4 Cell Count > 500: Group which contains naive patients with CD4 nadir more than 500 cell/mkl at the moment of enrollment
- CD4 Cell Count 350-500: Group which contains naive patients with CD4 nadir between 350 and 500 cell/mkl at the moment of enrollment
- CD4 Cell Count < 350: Group which contains naive patients with CD4 nadir less than 350 cell/mkl at the moment of enrollment
Arm/Group | CD4 Cell Count > 500 | CD4 Cell Count 350-500 | CD4 Cell Count < 350
Number analyzed (Participants) | 161 | 116 | 159
participants
  R5-tropic | 123 | 85 | 114
  X4-tropic | 38 | 31 | 45

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Naïve Patients, >500 | Naïve Patients, 350-500 | Naïve Patients, <350 | ARVT <6 Months | ARVT From 6 Months to 3 Years | ARVT >3 Years
Serious Adverse Events (participants affected / at risk) | 0/179 | 0/140 | 0/176 | 0/122 | 0/172 | 0/154
Other Adverse Events (participants affected / at risk) | 0/179 | 0/140 | 0/176 | 0/122 | 0/172 | 0/154

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes